CLINICAL TRIAL: NCT04175041
Title: A Dose-Response Study of the Cognitive and Physiological Effects of tDCS to the DLPFC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, Chief of Division of Neuropsychiatry, Director of TMS Clinic, Director of Lab for Neuropsychiatry and Neuromodulation, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2018P002889
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Transcranial Direct Current Stimulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ADHD (Other): Patients with ADHD.
  Interventions: Device: Transcranial Direct Current Stimulation
- Healthy Control (Other): Volunteers without Neuropsychiatric Disorders.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — In tDCS, electrodes are applied on the scalp to transmit direct current at low current amplitudes.

SUMMARY:
To determine the cognitive and neurophysiological dose-response relationships of anodal tDCS to the left DLPFC as a function of absolute current intensity, individualized E-field intensity, and stimulation duration.

DETAILED DESCRIPTION:
To determine the cognitive and neurophysiological dose-response relationships of anodal tDCS to the left DLPFC as a function of absolute current intensity, individualized E-field intensity, and stimulation duration.

ELIGIBILITY:
Inclusion Criteria (Patients)

1. Male and female outpatients 18-55 years of age
2. A diagnosis of ADD/ADHD or meeting the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
3. Patient will be either off stimulant medications or, if undergoing treatment with stimulants, will be asked to discontinue two days prior to the experiment, under physician-guided protocol, and allowed to resume afterwards. Subjects may resume stimulant use between the two study visits so long as they discontinue use two days prior to the second study visit. If fatigue is problematic in subjects discontinuing medication, they will be allowed to continue with the study if they are able to follow the suggested taper plan (50% of the dose day one, 25% dose day 2, stop day of visit (day 3)).
4. If on non-stimulant medications, dose must have been stable for at least 4 weeks.

Exclusion Criteria (Patients)

1. Contraindication to tDCS: history or epilepsy, metallic implants in the head and neck, brain stimulators, vagus nerve stimulators, VP shunt, pacemakers, pregnancy.
2. Active substance dependence (except for tobacco).
3. Pregnant or nursing females.
4. Inability to participate in testing procedures.

Inclusion Criteria (Healthy Control)

1. Male and female outpatients 18-55 years of age

Exclusion Criteria (Healthy Control)

1. Diagnosis of psychiatric of neurological disorder
2. Ongoing treatment with any psychotropic medications.
3. Contraindication to tDCS: history or epilepsy, metallic implants in the head and neck, brain stimulators, vagus nerve stimulators, VP shunt, pacemakers, pregnancy.
4. Active substance dependence (except for tobacco).
5. Pregnant or nursing females.
6. Inability to participate in testing procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Accuracy and Reaction Time in Attention and Working Memory | Change Before and After Stimulation on Each of the Four Visits, Average of 2-6 Weeks
  Measured using Eriksen Flanker Task (EFT)

SECONDARY OUTCOMES:
Amplitude of Electroencephalogram (EEG) Event Related Potentials | Change Before and After Stimulation on Each of the Four Visits, Average of 2-6 Weeks
  Measure of amplitude related to stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Joan Camprodon, MD, PhD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States